CLINICAL TRIAL: NCT02603627
Title: Cross-sectional Study to Compare the Prevalence of Chronic Obstructive Pulmonary Disease (COPD) in Patients Newly Diagnosed With Lung Cancer, Compared to Controls
Brief Title: Prevalence of COPD in Our Lung Cancer Population, Compared to Controls
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RJ115/N106; 15/YH/0091 (Other: Yorkshire and the Humber REC)
Record Dates: First submitted 2015-08-11; First posted 2015-11-13 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-10

CONDITIONS: COPD; Lung Cancer; Smoking
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms; Smoking

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- With lung cancer: Patients who have a new diagnosis of lung cancer will be invited to undergo spirometry to enable us to gather data on the prevalence of COPD in this group.
- Without lung cancer: Smokers who are referred to the smoking cessation clinic will be invited to undergo spirometry to ascertain the prevalence of COPD in this group.

SUMMARY:
This study will investigate the prevalence of chronic obstructive pulmonary disease (COPD) in patients who are newly diagnosed with lung cancer and compare it to the prevalence of COPD in controls recruited from a smoking cessation clinic.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a breathing problem that some people develop. Usually it is caused by smoking. Damage to the lungs means that patients are at risk of more chest infections and are unable to exercise like healthy individuals. They may also have a long-standing cough.

COPD is diagnosed by testing lung function, usually using a small device called a spirometer.

COPD is becoming a better understood condition. It is known that the lungs of patients with COPD are sometimes inflamed. This is important because inflammation is associated with some types of cancer, including lung cancer.

The investigators are interested in whether COPD puts people at higher risk of lung cancer. They would like to find out how common COPD is in patients who have lung cancer. The investigators would also like to find out how common COPD is in patients who are not known to have lung cancer (comparison group). This will help them interpret their results better as investigators will be able to compare the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Aged over 18
* Lung cancer group: new diagnosis of lung cancer, with spirometry results available Control group: spirometry result available or obtained

Exclusion Criteria:

* Patient refusal
* Age under 18
* Control group: pre-existing lung cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the multidisciplinary lung cancer clinic at Guy's Hospital.
  Controls will be recruited from the smoking cessation clinic at Guy's and St Thomas' NHS Foundation Trust.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of COPD in lung cancer compared to controls, using spirometry to diagnose COPD. | Up to nine months

SECONDARY OUTCOMES:
Comparison of the proportion of small cell tumours to non-small cell tumours in patients with lung cancer and COPD. | Up to nine months
  No change to routine care (no extra specimens to be taken or retained), but data on the histological subtypes will be recorded (as described above) to better inform the investigators about whether COPD-associated lung cancer demonstrates a different histological subtype.
Comparison of the proportion of individuals with an emphysematous phenotype to the proportion of individuals with a bronchitic phenotype. | Up to nine months
  No change to routine care (no extra investigations to be performed), but data on the radiological phenotype will be recorded to better inform the investigators about whether patients with COPD-associated lung cancer tend to have an emphysematous COPD pattern or a bronchitic one.

CONTACTS AND LOCATIONS:
Overall Officials: Tariq Sethi, MBBS PhD, Principal Investigator — King's Health Partners; Anthony Dorr, MBBS PhD, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, England, United Kingdom